CLINICAL TRIAL: NCT05604820
Title: The Effect of Progressive Muscle Relaxation Exercise on Sleep Quality in Cancer Patients Receiving Chemotherapy: A Randomized Controlled Study
Brief Title: The Effect of Progressive Muscle Relaxation Exercise on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: KARATAY.ebru.sari001
Record Dates: First submitted 2022-10-16; First posted 2022-11-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cancer Patients

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the characteristics of the study, blinding cannot be applied to the participants. In order to eliminate the bias, the data of the study will be collected and recorded by an impartial researcher (assistant researcher) who does not know the groups trained by the researcher. The statistics of the research will be carried out by an independent statistician who does not know the groups. In this way, the prevention of bias will be ensured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Progressive Muscle Relaxation Exercise
  Interventions: Behavioral: Progressive Muscle Relaxation Exercise
- no ıntervention (No Intervention)

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation Exercise — Training on progressive muscle relaxation exercises will be given to the experimental group in the chemotherapy unit. Before going to sleep in the evening and during the day, they will be asked to do progressive muscle relaxation exercises in line with the instruction of the video. They will be asked to do the application every day for 8 weeks. At the end of the 2nd week, 4th week, 6th week and 8th week, they will be asked to fill the PUKI again. Only routine care will be applied to the control group and no intervention will be made. At the end of the 2nd week, 4th week, 6th week and 8th week, they will be asked to fill the PUKI again. After the evaluations, information about progressive muscle relaxation exercises will be given.
  Arms: experimental

SUMMARY:
Chemotherapy is applied as a standard method in the treatment of cancer, which is an important public health problem in terms of incidence and mortality. Sleep quality due to cancer and its treatments is adversely affected. Cognitive behavioral therapies, walking and relaxation exercises are known to be beneficial in increasing sleep quality. For this reason, this study will be conducted to evaluate the effect of progressive muscle relaxation exercises applied to individuals who are undergoing chemotherapy and whose sleep quality has deteriorated, on sleep quality. The research will be carried out between March and September 2022 in Konya City Hospital Chemotherapy Unit with patients undergoing chemotherapy. Patients who will receive chemotherapy will be informed about the study, and those who accept to participate in the study will be evaluated according to the inclusion and exclusion criteria of the sample selection. They will be asked to fill out the PUKI. It will then be assigned to the control or experimental group with the randomization program assignment. Training on progressive muscle relaxation exercises will be given to the experimental group in the chemotherapy unit. Before going to sleep in the evening and during the day, they will be asked to do progressive muscle relaxation exercises in line with the instruction of the video. They will be asked to do the application every day for 8 weeks. At the end of the 2nd week, 4th week, 6th week and 8th week, they will be asked to fill the PUKI again. Only routine care will be applied to the control group and no intervention will be made. At the end of the 2nd week, 4th week, 6th week and 8th week, they will be asked to fill the PUKI again. After the evaluations, information about progressive muscle relaxation exercises will be given.

DETAILED DESCRIPTION:
Chemotherapy is defined as treatment with chemical drugs that prevent the proliferation of malignant tumor cells, kill the cell or stop its function. Since these chemical agents affect healthy cells as well as diseased cells, they can cause serious side effects . These side effects include nausea, vomiting, increased risk of infection due to bone marrow suppression,mucositis, insomnia, diarrhea, constipation, fatigue, organ toxicity such as cardiotoxicity, nephrotoxicity. . These conditions cause patients to be negatively affected physically and psychosocially. Prevention of these side effects that develop due to chemotherapy plays a role in the timely and effective dosing of chemotherapy.Sleep disorders, which negatively affect sleep quality, which is one of the side effects, are observed in 30-50% of cancer patients due to chemotherapy . In studies, sleep disorders and sleep quality negatively affect the quality of life by causing frequent cognitive disorders, inability to collect attention, daytime dysfunctions, fatigue. In addition, deterioration of sleep quality causes delay in wound healing, difficulty in performing daily activities, deterioration of clinical and treatment compliance . Progressive November Relaxation therapy is a mind-body technique that involves stretching slowly and is used to relieve stress. Relaxation can be quite beneficial if practiced routinely. Progressive muscle Relaxation November exercises are widely used by people to reduce anxiety and cope. November The principle of the Progressive Muscle Relaxation exercise is based on relaxation after November, when the muscles are strongly stretched. The patient is taught to be consciously sensitive to the body. In general, relaxation techniques include calming down, refocusing on something, and increasing physical awareness. Relaxation techniques, slowing heart rate and respiratory rate, reduce blood pressure, by increasing blood flow to many main group, Nov, Nov, reducing tension and chronic pain, together with the concentration of the individual increases. Relaxation-based treatment approaches are based on the conclusion that patients with sleep disorders often have excessive physiological and cognitive arousal day and night. Relaxation methods are used to disable the arousal system.Progressive muscle relaxation exercises are easy-to-learn exercises that do not cost anything and are thought to be effective in improving November sleep quality in patients receiving chemotherapy. For this purpose, this study was planned to evaluate the effect of progressive November relaxation exercises on sleep quality in patients receiving chemotherapy.The quality of sleep is that the individual feels rested, vigorous and ready for a new day. Sleep quality occupies an important place in clinical practice and sleep research. The reason for this is that individuals with low and poor sleep quality are more likely to encounter physiological and psychological health problems than individuals who sleep a quality sleep . There are many factors that affect sleep, sleep duration and sleep quality. These factors are often not related to a single factor, but sleep problems occur due to more than one reason physically, environmentally and psychologically. These reasons are diseases, environmental factors, age, gender, psychological factors, smoking, medications, nutrition, etc. they are factors.Since a quality and adequate sleep accelerates the recovery process of patients, sick individuals need more sleep and rest than healthy individuals. Nurses can determine whether the patient has sleep problems with the data they receive from the patient as the first source. In patients with sleep problems, they can apply nursing interventions for the sleep disorder experienced by the patient by evaluating the frequency and duration of this condition. By approaching sick and healthy individuals holistically, nurses can identify sleep problems and other needs that affect and may affect them in advance. And they can improve the sleep quality of patients and healthy individuals with PKG.Progressive November relaxation exercise is one of the cognitive-behavioral treatment techniques that allows voluntary contraction and relaxation of muscles. November relaxation is one of the most effective and effective methods of cognitive-behavioral therapy. The term progressive relaxation is a relative reduction in the severity of tension November seen in skeletal muscles. PKG is a type of muscle groups in the body (hand, arm, neck, shoulder, face, chest, abdomen, buttocks, legs, feet, November, etc.).) involves its stretching and relaxation. With this method, the application is started from the November muscles in the head-neck area and progressed to the feet. PKGE is one of the easy-to-learn, cost-free, practical and side-effect-free methods.This research is a randomized controlled trial in which the effect of progressive muscle relaxation exercises applied to individuals receiving chemotherapy for cancer on sleep quality was examined November.November February 10, 2022- February 20, 2023 The research will be conducted at the Chemotherapy Unit of Konya City Hospital. Dec. The Chemotherapy Unit is a unit with 39 seats and 5 rooms where outpatient chemotherapy applications for cancer treatment are performed. In the unit, two medical oncologists, nine oncology nurses and an oncology education nurse who provides training on side effects of chemotherapy are serving. The unit started to serve on July 2, 2021 and chemotherapy is administered to an average of 350 cancer patients per month, especially lung cancer and breast cancer. The average number of daily chemotherapy applications is 100. After deciding on chemotherapy treatment for patients who will undergo chemotherapy and creating a chemotherapy protocol, chemotherapy is administered in accordance with the chemotherapy protocol. Before applying chemotherapy, the oncology training nurse provides training on the drugs included in the chemotherapy protocol, the frequency of application, duration of application, possible side effects of chemotherapeutic drugs, as well as recommendations for what the patient and relatives should do about these possible side effects. Before applying chemotherapy, the patient is evaluated for vital signs and conditions that are contraindicated in chemotherapy, such as leukopenia, the presence of infection, and chemotherapy is administered to patients who do not have any problems applying chemotherapy. Chemotherapeutic drugs are prepared and administered at the chemotherapy preparation center located in the unit.The Universe and Sample of the Research The universe of the research will be composed of patients receiving chemotherapy in the chemotherapy unit where the research will be conducted. July Decembers 2021-December 2021 chemotherapy was administered to a total of 2100 patients in the chemotherapy unit. The number of samples was determined according to the results of a similar study using the G*Power 3.1.9.7 program with α = 0.05 and 80% power. 31 to 62 in each group is calculated as the number of participant sample, and by considering the potential losses during operation this number to 40 participants for each group was 80.

Criteria for Inclusion in the Study Pittsburgh Sleep Quality Index (PUKI) score, which is 5 points and above, who are 18 years of age or older, Who will receive outpatient chemotherapy in the chemotherapy unit, Knows how to read and write, Using mobile phone conveniently to upload progressive November relaxation exercise video, Who volunteered to participate in the research. Criteria for Non-Inclusion in the Study Hearing impaired, Receiving radiotherapy treatment, Who has a physical disability to perform relaxation exercises, Depression, schizophrenia, etc. with a diagnosis of psychiatric illness, With neurological disorders, With a metastatic condition, Antidepressants or sleeping pills, etc. using medication, Relaxation exercise (yoga, breathing and meditation, etc.) acting. Termination Criteria Who cannot perform relaxation exercises at least 2 days in a row and at least 9 days in a month during the research process, Chemotherapy treatment is terminated for any reason during the intervention Variables of the Research Independent Variable: Progressive November muscle relaxation exercises Dependent Variable: Sleep quality and sleep quality sub-dimensions (subjective sleep quality, sleep latency, habitual sleep efficiency, sleep disturbance, sleep medication use, and daytime dysfunction) Research Hypothesis H November 1: The total PKI score of patients who received chemotherapy and performed progressive muscle relaxation exercises is lower than the total PKI score of patients who did not perform progressive November relaxation exercises.

Collection of Data In this section, information about data collection tools will be given. Data Aggregate Tools In the research, the data will be collected using the Introductory Information Form, Pittsburgh

Pittsburgh sleep quality index :

Developed by Buysse et al., PUKI, which was validated and reliable in Turkish by Ağargün, is a self-reported assessment tool that provides information about the quality of sleep and the type and severity of sleep disorders in the last month. It consists of a total of 24 questions, including 19 questions that assess the quality, quantity, presence and severity of sleep disorders in an individual, and 5 questions answered by the individual's spouse or roommate.

Application of Research The implementation phase of the research is indicated in Table 1 and Figure 1. Randomization Randomizasyon.org groups from the site will be randomized by the block randomization method by a researcher who knows the research other than the researcher. The numbers in the randomization list will be placed in closed envelopes according to the order. Patients who meet the criteria for admission to the study will be assigned according to this list after their consent is obtained and preliminary tests are completed.

Blinding Due to the characteristics of the study, blinding cannot be applied to the participants. In order to eliminate the bias, the data of the study will be collected and recorded by an impartial researcher (assistant researcher) who does not know the groups trained by the researcher. The statistics of the research will be carried out by an independent statistician who does not know the groups. In this way, the prevention of bias will be ensured.

Statistical Evaluation of Research Data Statistical analysis of the data obtained as a result of the research will be carried out in IBM SPSS 25 (Statistical Package For Social Sciences) program. Number, percentage, standard deviation and arithmetic mean will be used as descriptive statistics in the analysis of the data. Parametric and nonparametric tests will be applied according to the normality test results. The results obtained will be tested at the p<0.05 significance level.

The Ethical Dimension of Research In order to conduct the research, the approval of the Ethics Committee of KTO Karatay University Interventional (Non-Invasive) Clinical Research Ethics Committee and the permission of the institution where the research will be conducted will be obtained. Volunteering is the basis for participation in the study and written consent will be obtained from the participants. (Additional. 9. Written Consent Form). Permission was obtained from Mehmet Ağargün for the Pittsburgh Sleep Quality Index (PUKI). (Additional. 6. Permission to use the Pittsburgh sleep quality index). Permission for use has been obtained from the Turkish Psychological Association for progressive November relaxation exercises CD. (Additional. 5. Progressive muscle relaxation exercise cd permission). November........... In order to prevent bias, Clinical Trials protocol registration will be made after obtaining permission from the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Pittsburgh Sleep Quality Index (PUKI) score, which is 5 points and above,

  * who are 18 years of age or older,

    * Who will receive outpatient chemotherapy in the chemotherapy unit,
  * Knows how to read and write,
  * Using mobile phone conveniently to upload progressive November relaxation exercise video, * Who volunteered to participate in the research.

Exclusion Criteria:

* * Hearing impaired,

  * Receiving radiotherapy treatment,
  * Who has a physical disability to perform relaxation exercises,
  * Depression, schizophrenia, etc. with a diagnosis of psychiatric illness,
  * With neurological disorders,
  * With a metastatic condition,
  * Antidepressants or sleeping pills, etc. using medication,
  * Relaxation exercise (yoga, breathing and meditation, etc.) acting.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
quality of sleep | two months
  measuring the effect of progressive November relaxation exercise on sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Kto Karatay üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No